CLINICAL TRIAL: NCT00531375
Title: The Effect of Silicone Hydrogel Contact Lenses on Conjunctival Flora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Clinical Vision Research Australia (Other); Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Dr Carol Lakkis, Clinical Vision Research Australia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H07 003
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Device: Silicone hydrogel contact lens

SUMMARY:
The primary purpose of this study is to investigate the effect of silicone hydrogel contact lenses on conjunctival flora over a period of 6 months of daily wear. A secondary aim is to compare the levels of microbial contamination of silicone hydrogel lenses after daily wear.

ELIGIBILITY:
Inclusion Criteria:

* Is correctable to at least 6/9 distance visual acuity in each eye with spherical contact lenses.
* Is a current full time soft contact lens wearer.
* Has no clinically significant anterior eye findings.
* Has no other active ocular disease

Exclusion Criteria:

* Has any systemic disease that might interfere with contact lens wear
* Is using any systemic or topical medications that will affect ocular health.
* Has any pre-existing ocular irritation that would preclude contact lens fitting.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (dry eyes) that would affect the wearing of contact lenses.
* Has undergone corneal refractive surgery.
* Is pregnant, lactating or planning a pregnancy.
* Is participating in a concurrent clinical trial.
* Has a latex sensitivity.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lakkis, BScOptom, PhD, PGCertOcTher, Principal Investigator — Clinical Vision Research Australia, Victorian College of Optometry
Locations (1):
- Clinical Vision Research Australia, Melbourne, Victoria, Australia